CLINICAL TRIAL: NCT05469191
Title: Effect of the Sit to Stand Test on Muscle Architecture After Eight Weeks.
Brief Title: Eight-week Effect of the Sit-to-stand Test on Muscle Architecture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Rodrigo Lizama Perez, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IDAFISAD 64201
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Quality Muscle; Arquitecture Muscle

STUDY DESIGN:
Intervention Model Description: A group that will perform the 5 STS will be compared with a group that will perform the 10 STS for 8 weeks, and there will also be a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 5 STS (Experimental): Group 5 STS will perform the same protocol as group 10 STS, only the number of repetitions between each set will change.
  Interventions: Other: Group 5 STS
- Group 10 STS (Experimental): Group 10 STS will perform the same protocol as group 5 STS, only the number of repetitions between each set will change.
  Interventions: Other: Group 10 STS
- Control group (No Intervention): Control group, no intervention.

INTERVENTIONS:
Other: Group 5 STS — For 8 weeks, 3 times per week and 3 sets of 5 repetitions during the first month, then 5 sets of 5 repetitions during the second month.
  Between each repetition, there will be a rest of 30 to 60 seconds approximately.
  Arms: Group 5 STS
Other: Group 10 STS — For 8 weeks, 3 times per week and 3 sets of 10 repetitions during the first month, then 5 sets of 10 repetitions during the second month.
  Between each repetition, there will be a rest of 30 to 60 seconds approximately.
  Arms: Group 10 STS

SUMMARY:
An 8-week intervention of the sit-to-stand test (STS) of 5 and 10 repetitions will be performed to two randomly selected groups to compare its effect on the muscle architecture of the vastus lateralis muscle.

H1: 10 STS significantly modifies vastus lateralis muscle architecture in adults compared to 5STS and the control group.

DETAILED DESCRIPTION:
Participants will be required to attend the laboratory for a first familiarization visit, where descriptive, biometric, and medical variables will also be evaluated. In addition, during this first familiarization session, it will be previously determined if the participants present any exclusion criteria and their muscle architecture will also be evaluated. After the familiarization session and the participants have signed the informed consent form, they will be randomly assigned to a 5 STS, 10 STS, or control group. Each group (exception of the control group) will be asked to perform three times a week one of the STS modalities assigned to them for 8 weeks, to ensure that the test is completed correctly and also to maintain the planning, the evaluator will be connected virtually with the participants, where rest times will be controlled and a fatigue perception scale will be performed at the end of each session, which will allow controlling the process each session. Subsequently, participants will be asked to attend the laboratory to re-evaluate their architectural parameters ( pennation angle, fascicle length, and muscle thickness) of the quadriceps muscle, one week after performing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over 18 years of age.
* They must have signed the informed consent form.
* Who can perform the STS.
* In case of suffering from a chronic non-communicable disease, that it is under control.

Exclusion Criteria:

* Inability to perform the STS.
* Hypertension (>200/110 mmHg).
* Acute neuromuscular or joint injury.
* Who have suffered a stroke in the last 6 months.
* Who have suffered a myocardial infarction or fracture in the last 6 months.
* Terminally ill.
* People who practice a sport professionally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change in the pennation angle of the vastus lateralis muscle. | Before, 1 week completion of the intervention.
  Calculated as the angle of insertion of the muscle fiber fascicles into the deep aponeurosis, measured with a linear probe in B-mode.
Change in the length of the fascicle of the vastus lateralis muscle | Before, 1 week after completion of the intervention.
  is calculated by measuring the length of the fascicular pathway between the superficial and deep aponeuroses,measured with a linear probe in B-mode.
Change in vastus lateralis muscle thickness | Before, 1 week after completion of the intervention.
  Muscle thickness will be determined as the distance between the superficial aponeurosis to the deep aponeurosis, measured with a linear probe in B-mode.
Change in muscle quality index (MQI) | Before, 1 week after completion of the intervention.
  Was calculated using two different formulas: one proposed by Takai et al. And one by Fragala et al. The "Takai formula" considers the time required to perform ten repetitions of the sit-to-stand test, while the "Fragala formula" uses the time required for five repetitions: MQI = ((leg length x chair height) x body mass x gravity x 10/ Time STS). Both calculations consider the length of the leg in meters, the height of the chair used in the test, body mass in kilograms, acceleration due to gravity (9.81 m/s^2), and a fixed constant of 10.

SECONDARY OUTCOMES:
Change in STS mean velocity (m· s-1), STS mean force (N), STS mean power (W), and STS relative power (W·Kg-1) | Before, 1 week after completion of the intervention.
  The STS mean velocity (m· s-1), STS mean force (N), STS mean power (W), and STS relative power (W·Kg-1), were calculated with the formulas proposed by Alcazar et al. The formulas are as follows:
  1. STS mean velocity = [0.5 x Height - Chair height] / Five STS time × 0.1]
  2. STS mean force = 0.9 x g x Body mass
  3. STS mean power = Body mass x 0.9 x g x [Height x 0.5 - Chair height / Five STS time × 0.1]
  4. Relative STS mean power = 0.9 x g x Height [ 0.5 x Chair height] / Five STS time × 0.1]

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Lizama Pérez, M.Sc, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad San Sebastián, sede Valdivia., Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No